CLINICAL TRIAL: NCT06371482
Title: Durvalumab Combined With Chemoradiotherapy for Limited Stage Small Cell Lung Cancer
Brief Title: Durvalumab Combined With Chemoradiotherapy for Limited Stage Small Cell Lung Cancer (Camel-01)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Camel-01
Record Dates: First submitted 2024-03-27; First posted 2024-04-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-03

CONDITIONS: SCLC, Limited Stage
Keywords: SCLC, Limited Stage; immunotherapy; chemoradiotherapy; Durvalumab
MeSH Terms: interventions — durvalumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- D with CRT (Experimental): The patients with limited stage small cell lung cancer receive durvalumab combined with chemoradiotherapy.
  Interventions: Drug: Durvalumab; Drug: Chemotherapy drug of EP regimen; Radiation: radiotherapy

INTERVENTIONS:
Drug: Durvalumab — Durvalumab is an immunoglobulin G (IgG) 1-κsubtype monoclonal antibody (mAb) that blocks the interaction of PD-L1 with PD-1 in T cells and CD80 (B7.1) in immune cells (ics). Durvalumab is developed by Astrazeneca /MedImmune for the treatment of cancer. Durvalumab is designed to reduce the cytotoxicity of antibody-dependent cells and complement dependent cytotoxicity. In vitro studies have demonstrated that Durvalumab can antagonize the inhibition of PD-L1 in human primary T cells, causing them to resume proliferation and release interferon gamma (IFNγ). To date, more than 1,800 patients have been treated with valiuzumab as a single agent or in combination with other cancer agents as part of ongoing studies. Durvalumab: 10mg/Kg, intravenously, starting at week 7 every 3 weeks for at least 1 year, or until progression, intolerance, or spontaneous withdrawal of the patient.
Drug: Chemotherapy drug of EP regimen — Etoposide: 80-100mg/m², intravenous infusion, given at week 1, 4, 7, 10, 13, 16, a total of 6 cycles.
  Carboplatin: AUC=5-6, intravenous infusion, given at weeks 1, 4, 7, 10, 13, 16, a total of 6 weeks. Or cisplatin: 75-80mg/m2 intravenously, given at weeks 1, 4, 7, 10, 13, 16 for a total of 6 weeks.
Radiation: radiotherapy — Radiotherapy: Total dose of 60Gy/30 times, each time 2.0Gy, 5 times a week from week 7 to week 12 of radiotherapy.

SUMMARY:
This trial aims to assess efficacy and safety of durvalumab combined with chemoradiotherapy for limited stage small cell lung cancer.

DETAILED DESCRIPTION:
Small cell lung cancer is a highly malignant tumor that accounts for about 15% of all lung cancer types. The 5-year survival rate is less than 5%, and the overall survival of patients who do not receive any antitumor therapy is only 2-4 months. In the past 40 years, 4 to 6 cycles of platinum-based chemotherapy, that is, etoposide combined with cisplatin or carboplatin, has become the standard therapy for small cell lung cancer patients and has been recommended by major global tumor treatment guidelines. While initial response rates are as high as 70%, 80% of limited-stage patients and nearly all patients with extensive stages are found to experience relapse or disease progression. Current guidelines recommend that patients with limited stage small cell lung cancer adopt the EP regimen combined with thoracic radiotherapy as the preferred treatment for patients with limited stage small cell lung cancer. PD-L1 is part of a complex system of receptors and ligands involved in controlling T cell activation. PD-L1 acts at multiple sites in the body, releasing inhibitory signals to T cells via the PD-1 and CD80 receptors to help regulate the immune response. Durvalumab is an immunoglobulin G (IgG) 1-κsubtype monoclonal antibody (mAb) that blocks the interaction of PD-L1 with PD-1 in T cells and CD80 (B7.1) in immune cells (ics). This trial aims to assess efficacy and safety of durvalumab combined with chemoradiotherapy for limited stage small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation and written signed informed consent;
* Age 18-75 years old, gender is not limited;
* Histologically or cytologically confirmed limited-stage small cell lung cancer (2009 AJCC/UICC/IASLC lung cancer TNM staging criteria, limited-stage SCLC is any T stage, any N stage, and M0), and patients with suspected brain or bone metastasis at the time of screening should undergo brain MRI or ECT before study enrollment;
* There are immunohistochemical results;
* Chemotherapy must include either cisplatin or carboplatin, in combination with etoposide;
* Physical status score ECOG 0-1;
* Weight > 40 kg;
* Expected survival ≥ 6 months;
* According to RECIST 1.1 guidelines, at least one lesion (not previously receiving radiotherapy) with a maximum diameter ≥ 10 mm as accurately measured by computed tomography (CT) or magnetic resonance imaging (MRI) at baseline (except lymph nodes, whose short axis must be ≥ 15 mm); And the lesion is suitable for repeated accurate measurement.;
* No previous immunotherapy;
* no serious abnormalities of haematopoietic, cardiac, pulmonary, hepatic; and renal functions and immunodeficiency (Haematology: white blood cells ≥3.5×109/L; neutrophils ≥1.5×109/L; haemoglobin ≥90g/L; platelets

  ≥100×109/L. Liver and kidney function: total bilirubin ≤1.5 times the upper limit of normal (ULN); AST (SGOT) and ALT (SGPT) ≤2.5 times the upper limit of normal; creatinine ≤1.5 times the upper limit of normal; albumin ≥30 g/L. Coagulation: International Normalised Ratio (INR) or Prothrombin Time (PT) or Activated Partial Thromboplastin Time (APTT)

  ≤ 1.5 times ULN; if the subject is receiving anticoagulation therapy, PT or INR is acceptable as long as the PT or INR is within the range of the anticoagulant drug formulation. Echocardiographic assessment: left ventricular ejection fraction (LVEF) ≥ low limit of normal (50%). Pulmonary function FEV1 ≥70% of % of predicted value and DLCO ≥60% of % of predicted value).
* The female patient has evidence of postmenopausal status, or the urine or serum pregnancy test results of the premenopausal woman are negative. Women who stop menstruating for 12 months without other medical reasons are considered menopausal.

Exclusion Criteria:

* Distant organ metastases (excluding supraclavicular lymph nodes) as determined by CT evaluation during screening and prior imaging;
* have received prior radiotherapy to the chest;
* have medical contraindications to etoposide - platinum (carboplatin or cisplatin) based chemotherapy;
* having any active autoimmune disease or a history of autoimmune disease (e.g. interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary gland inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (which can be included if hormone replacement therapy is effective), etc.), and a history of immunosuppressive drug use within 28 days, with the exception of the use of hormones for the purpose of dealing with toxicity from radiotherapy;
* Previously received or are receiving other PD-1 antibody therapy or other immunotherapy targeting PD-1/PD-L1, or are currently participating in other interventional clinical studies for treatment;
* Have received other anti-tumour therapy (including herbal therapy with anti-tumour effect) within 4 weeks prior to the first dose of the study; have received long-term systemic immunotherapy or hormone therapy (except physiological replacement therapy, e.g., oral thyroxine for hypothyroidism) within 4 weeks prior to the first dose of the study; and have been treated with other experimental drugs or interventional clinical studies within 4 weeks prior to the first dose of the study;
* Patients with uncontrolled clinical cardiac symptoms or disease such as

  (1) NYHA class II or higher heart failure, (2) unstable angina pectoris, (3) myocardial infarction within 1 year, and (4) clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention;
* with congenital or acquired immune function defects (e.g., HIV-infected patients), active hepatitis B (HBV-DNA ≥104 copies/ml) or hepatitis C (hepatitis C antibody-positive with HCV-RNA above the lower limit of detection of the analytical method), or active tuberculosis;
* Have an active infection or unexplained fever >38.5°C within 2 weeks prior to screening (at the investigator's discretion, subjects may be enrolled for fever arising from tumours);
* In the judgement of the investigator, the subject has other factors that may cause him/her to be forced to terminate the study in the middle of the study, e.g., suffering from other serious illnesses (including psychiatric illnesses) that require comorbid treatment, family or social factors that may affect the safety of the subject or the collection of trial data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of objective remission rate (ORR) in limited stage small cell lung cancer treated with durvalumab combined with chemoradiotherapy | Treatment with durvalumab for at least 1 year, or until progression, intolerance, or spontaneous withdrawal of patients.
  Objective tumor remission is assessed by the investigator using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria). Objective remission rate (ORR): defined as the proportion of subjects whose tumor volume shrinks to a pre-specified value and can be maintained for the minimum time frame required, incorporating cases in complete remission (CR) and partial remission (PR).
Assessment of the incidence of treatment-related adverse events Incidence of Treatment-Emergent Adverse Events. | Treatment with durvalumab for at least 1 year, or until progression, intolerance, or spontaneous withdrawal of patients.
  Adverse events are observed during the course of the study and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE V5.0).

SECONDARY OUTCOMES:
Assessment of overall survival (OS) in limited stage small cell lung cancer. | Treatment with durvalumab for at least 1 year, or until progression, intolerance, or spontaneous withdrawal of patients.
  Objective tumor remission is assessed by the investigator using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria). OS is defined as the time from the start of enrollment to death from any cause.
Assessment of progression-free survival (PFS) in limited stage small cell lung cancer. | Treatment with durvalumab for at least 1 year, or until progression, intolerance, or spontaneous withdrawal of patients.
  Objective tumor remission is assessed by the investigator using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria). PFS is defined as the time from the start of enrollment until tumor progression or death from any cause.
Assessment of disease control rate (DCR) in limited stage small cell lung cancer. | Treatment with durvalumab for at least 1 year, or until progression, intolerance, or spontaneous withdrawal of patients.
  Objective tumor remission is assessed by the investigator using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria). Disease control rate (DCR): the proportion of patients whose tumors shrank or were stable and remained so for a certain period of time, including complete remission (CR), partial remission (PR) and stable disease (SD).

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Shen, PhD, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China